CLINICAL TRIAL: NCT04557969
Title: Prospective Study of Surgery in Gastrointestinal Stromal Tumors (GISTs) for Treatment, Tumor Modeling, and Genomic Analysis
Brief Title: Surgery in Gastrointestinal Stromal Tumors (GISTs) for Treatment, Tumor Modeling, and Genomic Analysis
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200161; 20-C-0161
Record Dates: First submitted 2020-09-18; First posted 2020-09-22 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-09-10

CONDITIONS: Gastric Cancer; Gastric Neoplasm; Gastrointestinal Stromal Sarcoma; Gastrointestinal Stromal Neoplasm; Gastrointestinal Stromal Tumor (GIST)
Keywords: Tyrosine Kinase Inhibitor (TKI) Therapy; Wild-Type GISTs (WT GISTs); PDGFRA Mutation; KIT Mutation; SDH Mutation; Natural History
MeSH Terms: conditions — Stomach Neoplasms; Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/ Cohort 1: Patients with histologically confirmed or clinical presentation suspicious of GIST

SUMMARY:
Objective:

To follow people with GISTs and collect tumor tissue so that it can be studied in the lab.

Eligibility:

People age 6 and older who have a GIST.

Design:

Participants will be screened with a review of their medical records and samples.

Participants will enroll in 1 other NIH study, and may be asked to enroll in 2 other optional NIH studies.

Participants will have a medical history and physical exam. Data about how they function in their daily activities will be obtained.

Participants may speak with a genetic counselor. They may have genetic testing.

Participants will give blood samples. They may have a cheek swab. For this, small brush will be rubbed against the inside of the cheek.

Participants may have a computed tomography (CT) scan of the chest, abdomen, and pelvis. Or they may have a CT scan of the chest and magnetic resonance imaging (MRI) of the abdomen and pelvis.

Participants will be monitored every 6-12 months at the NIH Clinical Center, for up to 10 years before having surgery. If they need surgery, it will be performed at the NIH. Then, they will be monitored every 6-12 months, for up to 5 years after surgery.

If a participant has surgery, tumor tissue samples and research specimen will be taken.

If a participant does not need surgery, their participation will end after 10 years. If they have surgery, the 5-year monitoring period will restart after each surgery.

DETAILED DESCRIPTION:
Background:

Gastrointestinal stromal tumors (GISTs) are the most common gastrointestinal soft tissue sarcoma, but remain a rare disease entity.

Most GISTs are characterized by KIT or PDGFRA mutations, making them susceptible to tyrosine kinase inhibitor (TKI) therapy.

Wild-type (WT) GISTs are rarer tumors, usually characterized by SDH mutations and/or lack of KIT or PDGFRA mutations; paragangliomas are frequently associated with WT GISTs.

Non-WT GISTs may become refractory to TKI therapy, whereas WT GISTs are generally resistant to TKI therapy.

The primary treatment modality for GISTs is surgical resection, which may involve the stomach, liver, and/or peritoneal surfaces; most patients will require multiple operations to remove disease not responsive to systemic agents.

Investigational systemic therapies are limited by toxicity and/or lack of efficacy, resulting in an unmet need for novel treatment options.

Obtaining fresh tumor tissue is critical to the successful development of GIST models for drug research, as well as for next generation tumor genomic sequencing, and to help identify novel targets and/or agents for the treatment of WT and TKI-resistant non-WT GISTs.

Objective:

Evaluate and follow participants with GISTs, particularly WT and treatment-refractory non-WT, to support translational research for this rare disease

Assess disease-free intervals (DFIs) between surgical resection of disease for at least 5 years

Eligibility:

Participants with histologically confirmed or clinical presentation suspicious of GIST.

Design:

Prospective cohort study

Participants with histologically confirmed or clinical presentation suspicious of GIST will enroll on study and will have active surveillance every 9-15 months for up to 10 years prior to and up to 5 years after surgical resection and/or cytoreduction. As participants may have multiple resections during the course of the study, 5-year surveillance post-surgery may be initiated multiple times, relative to the last resection performed.

All participants enrolled will be evaluated for tumor resection or cytoreduction at the start of study and if appropriate, will be offered surgery, otherwise they will be on active surveillance until surgical resection or cytoreduction is clinically indicated.

It is expected that approximately 30-40 participants per year may enroll on this trial; the accrual ceiling will be set at 400 to permit accrual over a 10-year period.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histological confirmation or clinical presentation suspicious of GIST; histological confirmation will be preferably by review of archival tissue if available, fresh biopsy will not be required if inadequate tissue sample.
* Age >= 6 years
* ECOG performance status <= 2 (Karnofsky or Lansky >= 60%)
* Ability of participant or parent/guardian to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

- Non-modifiable medical comorbidities that would preclude cytoreductive surgery.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with histologically confirmed or clinical presentation suspicious of GIST.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2040-12-30 (Estimated); Study Completion 2040-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate and follow patients with GISTs, particularly WT or treatment-refractory non-WT, to support translational research for this rare disease | on-going
  Patients with non-WT GIST and WT GIST will have the durations of the DFIs described both within each patient as their own control and across patients. Analyses will be done separately for those with WT GIST and those with non-WT GIST as well as for all patients combined.
Assess disease-free intervals (DFIs) between surgical resection of disease for at least 5 years | surveillance every 6-12 months and time of surgery, until 5 years after last surgical resection (relative to the last resection performed)
  Surveillance every 6-12 months and time of surgery, by tumor measurement and imaging studies, to assess disease-free intervals (DFIs) between surgical resection of disease for at least 5 years.

SECONDARY OUTCOMES:
Characterize genomic and clinicopathologic features of GISTs | at clinical visits and follow-up
  Characterization of the genomic and clinicopathologic features associated with GISTs.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Blakely, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-C-0161.html